CLINICAL TRIAL: NCT04330963
Title: International Swiss Primary Hypersomnolence and Narcolepsy Cohort Study
Acronym: iSPHYNCS
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Klinik Barmelweid (Other); Zentrum für Schlafmedizin Basel (Unknown); Ospedale Regionale di Lugano (Other); Cantonal Hospital of St. Gallen (Other); Zurzach Care Klinik für Schlafmedizin (Unknown); University Children's Hospital, Zurich (Other); University Children's Hospital Basel (Other); Centre Lausannios de Sommeil (Unknown); Private Universität Witten-Herdecke and Orfea Fachklinik für Schlafmedizin, Witten, Germany (Unknown); Leiden University Medical Center, Leiden, Netherlands (Unknown); University of Bologna, Bologna, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-00788
Record Dates: First submitted 2020-01-06; First posted 2020-04-02 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Narcolepsy; Idiopathic Hypersomnia; Hypersomnolence Disorder
MeSH Terms: conditions — Narcolepsy; Idiopathic Hypersomnia; Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Blood cerebrospinal fluid (CSF) Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hypersomnolence group: All patients referred to the outpatient clinic/sleep center for investigation due to complaints for excessive daytime sleepiness (EDS) and/or Hypersomnia (H) and/or suspected central disorder of hypersomnolence (CDH)
- Healthy controls: Healthy control subjects without complaints of EDS and /or H.
- SDB controls: Patients with EDS and diagnosis of severe sleep related breathing disorder (SBD) significantly improving with therapy.
- Pediatric Hypersomnolence group: Pediatric group aged 10-18. Same criteria for inclusion and exclusion apply as for the adult group.

SUMMARY:
Swiss Primary Hypersomnolence and Narcolepsy Cohort Study (SPHYNCS) is a cohort study on disease presentation and long-term course with an exploratory approach to detect biomarkers.

DETAILED DESCRIPTION:
An exploratory prospective, national, multi-center cohort study on clinical, electrophysiological and biological biomarkers of disease presentation and course.

ELIGIBILITY:
Inclusion Criteria:

Study participants:

* Subjective complaints of Excessive daytime sleepiness (EDS) and/or Hypersomnia (H) as defined above
* EDS and/or H present daily or almost daily for at least 1 month prior to the consultation
* Ability and consent to undergo electrophysiological routine assessment
* Ability to give informed consent

Healthy controls:

* Age and gender matched healthy subjects
* Including blood related relatives of study participants
* Ability and consent to undergo electrophysiological routine assessment
* Ability to give informed consent

Controls with Sleep disordered breathing (SDB):

* Subjective complaints of EDS with Epworth Sleepiness Scale (ESS) > 10 (adults) and/or H due to SDB: Presence of clinically significant and untreated obstructive sleep apnea (OSA) as determined by the investigator with an apnea-hypopnea-index >30/h
* Multiple sleep-latency test (MSLT) mean sleep latency ≤ 8min
* Subjective and objective improvement of EDS and/or H within 3 months after treatment with
* Positive airway pressure (PAP) therapy with documented

  * Reduction of apnea-hypopnea index below <10/h
  * Reduction of ESS by ≥ 25%
  * MSLT mean Sleep Latency > 12min
* Ability and consent to undergo electrophysiological routine assessment
* Ability to give informed consent

Exclusion Criteria:

Study participants and controls:

* SDB for study participants and healthy controls: Presence of clinically significant and untreated obstructive sleep apnea (OSA) or central sleep apnea (CSA) as determined by the investigator or documented previously; or documentation of one of the following:

  * Apnea index (AI) > 10 if on OSA treatment or untreated; or
  * Clinically significant hypoventilation; or
  * Noncompliance with primary OSA therapy
  * except if NT1 has been diagnosed including decreased or missing cerebrospinal fluid (CSF) hypocretin
* SDB for control population with SDB:

  * Central Sleep Apnea (CSA)
  * Noncompliance with primary OSA therapy and/or
  * No reported improvement of EDS and/or H within 3 months of positive airway pressure (PAP) treatment
* The following disorders/conditions that on clinical grounds are considered to be the cause of EDS / H

  * Other sleep disorders (e.g. Restless legs syndrome (RLS) with periodic leg movement syndrome (PLMS), sleepwalking, clear-cut circadian disorder)
  * Other neurological disorders (e.g. stroke, multiple sclerosis, parkinsonism, severe traumatic brain injury)
  * (Auto-)immune and systemic disorders (such as Hashimoto Thyroiditis, Chron's Disease, ulcerous colitis, Diabetes mellitus type I, Systemic lupus erythematosus)
  * Malignancy (except: Status in Remission for at least > 10 years)
  * Instable psychiatric disorder (e.g. acute psychotic, acute suicidal, episode of major depression requiring in-hospital treatment, active substance abuse)
  * Active infectious disease at screening
  * Permanent medications / drugs
* Chronic infectious diseases (such as Hepatitis B/C, HIV)
* Chronic use of antibiotics
* Recent use (< 8 weeks) of immune-modulating drugs

Healthy controls additional:

* Subjective complaints of EDS and / or H
* ESS > 10
* Polysomnography (PSG) with AI > 10/h and / or PLMS Index > 30/h
* MSLT mean Sleep Latency < 12 min

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The project population consists of subjects, who were referred to the outpatient clinic / sleep center of one of the study sites for further investigation, due to complaints of EDS and / or H and / or suspected Central disorders of hypersomnolence (CDH), fulfilling inclusion / exclusion criteria and a control population as well as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of study subjects with diagnosis of Narcolepsy type 1 (NT1) at follow up | 36 months
Proportion of study subjects with final diagnosis other than NT1 but within the group of CDH at follow up | 36 months

SECONDARY OUTCOMES:
Proportion of patients with autoreactive T-cell clones in NT1 and some Narcolepsy borderland (NBL) subjects but not in controls | 36 months
Preptidomic profile of NT1 and NBL in comparison to controls | 36 months
  Mass spectrometry based peptidomics of cerebrospinal fluid (CSF) for the identification of Hypocretin and approximately 6000 other neuropeptides in 10 to 20 samples for each group to be analyzed. In collaboration with the group of Prof. Matthias Mann, Max Planck Institute of Biochemistry, Planegg, Germany
Gut microbiome of NT1 and NBL in comparison to controls | 36 months
  16S based analysis of the gut microbiome based on stool samples from all participants (where available). In collaboration with the group of Prof. Andrew Macpherson, University of Bern

CONTACTS AND LOCATIONS:
Overall Officials: Claudio L Bassetti, Prof., Study Director — Insel Gruppe
Locations (1):
- Claudio L Bassetti, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassetti CLA, Adamantidis A, Burdakov D, Han F, Gay S, Kallweit U, Khatami R, Koning F, Kornum BR, Lammers GJ, Liblau RS, Luppi PH, Mayer G, Pollmacher T, Sakurai T, Sallusto F, Scammell TE, Tafti M, Dauvilliers Y. Narcolepsy - clinical spectrum, aetiopathophysiology, diagnosis and treatment. Nat Rev Neurol. 2019 Sep;15(9):519-539. doi: 10.1038/s41582-019-0226-9. Epub 2019 Jul 19. PMID 31324898
- [Background] Latorre D, Kallweit U, Armentani E, Foglierini M, Mele F, Cassotta A, Jovic S, Jarrossay D, Mathis J, Zellini F, Becher B, Lanzavecchia A, Khatami R, Manconi M, Tafti M, Bassetti CL, Sallusto F. T cells in patients with narcolepsy target self-antigens of hypocretin neurons. Nature. 2018 Oct;562(7725):63-68. doi: 10.1038/s41586-018-0540-1. Epub 2018 Sep 19. PMID 30232458
- [Background] Bassetti C, Aldrich MS. Idiopathic hypersomnia. A series of 42 patients. Brain. 1997 Aug;120 ( Pt 8):1423-35. doi: 10.1093/brain/120.8.1423. PMID 9278632
- [Background] Dietmann A, Wenz E, van der Meer J, Ringli M, Warncke JD, Edwards E, Schmidt MH, Bernasconi CA, Nirkko A, Strub M, Miano S, Manconi M, Acker J, von Manitius S, Baumann CR, Valko PO, Yilmaz B, Brunner AD, Tzovara A, Zhang Z, Largiader CR, Tafti M, Latorre D, Sallusto F, Khatami R, Bassetti CLA. The Swiss Primary Hypersomnolence and Narcolepsy Cohort study (SPHYNCS): Study protocol for a prospective, multicentre cohort observational study. J Sleep Res. 2021 Oct;30(5):e13296. doi: 10.1111/jsr.13296. Epub 2021 Apr 4. PMID 33813771
- [Derived] Morand R, Fregolente L, van der Meer J, Wenz ES, Helmy A, Brigato L, Warncke JD, Zub K, Khatami R, Zhang Z, von Manitius S, Miano S, Acker J, Strub M, Kallweit U, Lammers GJ, Tzovara A, Bassetti CLA, Mougiakakou S, Schmidt MH. iSPHYNCS: Unsupervised Clustering in Questionnaires and Metadata Reveals Distinct Subtypes in the Narcolepsy Borderland. J Sleep Res. 2026 Feb 9:e70294. doi: 10.1111/jsr.70294. Online ahead of print. PMID 41657285